CLINICAL TRIAL: NCT06360237
Title: Olezarsen (ISIS 678354) Early Access Program for Patients With Familial Chylomicronemia Syndrome (FCS)
Brief Title: Olezarsen Early Access Program for Patients With Familial Chylomicronemia Syndrome (FCS)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISIS 678354
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Familial Chylomicronemia Syndrome
Keywords: Familial Chylomicronemia; Familial Lipoprotein Lipase Deficiency; Hyperlipoproteinemias; Familial Hyperlipoproteinemia Type 1; Hyperlipoproteinemia Type 1; Hyperchylomicronemia, Familial; Lipoprotein Lipase Deficiency, Familial; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Lipid Metabolism, Inborn Errors; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome; Hyperlipoproteinemia Type I; Hyperlipoproteinemias; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Lipid Metabolism, Inborn Errors; Metabolic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn | interventions — olezarsen

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Olezarsen — Olezarsen 80 mg administered once monthly by subcutaneous (SC) injections in the abdomen, thigh, or upper arm.
  Other Names: ISIS-678354

SUMMARY:
The purpose of the Expanded Access Program is to provide pre-approval access of olezarsen to eligible patients with Familial Chylomicronemia Syndrome (FCS).

DETAILED DESCRIPTION:
The Expanded Access Program (EAP) is intended to provide pre-approval access to olezarsen for eligible patients with FCS who have limited or no available treatment options. This program is open in the United States and operates under the individual patient (also referred to as single patient) IND expanded access route in which the patient's treating physician serves as the sponsor. Expanded access requests must be from the patient's treating physicians and submitted according to the instructions at https://www.ionispharma.com/patients/expanded-access-policy/

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of FCS as determined by the sponsoring physician. Ionis will review each application to determine eligibility based on documentation of validated genetic or clinical diagnosis.

  o Documented loss of function mutations (homozygous, compound / double heterozygous) in genes such as LPL, GPIHBP1, APOA5, APOC2 or LMF1) or clinically validated diagnosis of FCS.
* Resides in and is a resident of the United States.
* Willing to follow a diet comprising ≤20 g fat per day.

Exclusion Criteria:

* Has any new or worsening of existing conditions which, in the opinion of the physician, would make the patient unsuitable for treatment with olezarsen.
* Olezarsen naïve patients with baseline platelet count <100x109/L at qualification.
* Estimated GFR (eGFR) <30 mL/min/1.73 m2.
* Secondary factors are the cause of triglyceride elevations.
* Is currently hospitalized in an acute emergency setting.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Expanded Access Site, Carlsbad, California, United States

REFERENCES:
- See also: Related Info — https://www.ionispharma.com/patients/expanded-access-policy/